CLINICAL TRIAL: NCT01797484
Title: Reduction of Ischemic Myocardium With Ranolazine-Treatment in Patients With Acute Myocardial Ischemia
Acronym: RIMINI-Pilot
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Tjark Frederik Schwemer, Dr. med., Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHZ-KARD-01-2013
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Results first posted 2018-01-12 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Coronary Artery Disease; Acute Myocardial Ischemia
Keywords: ischemia; myocardium; Ranolazine; dyskinesia; speckle tracking echocardiography
MeSH Terms: conditions — Coronary Artery Disease; Ischemia; Dyskinesias | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranolazine (Active Comparator): Ranolazine 500mg bid orally 7 days Ranolazine 750mg bid orally 35 days
  Interventions: Drug: Ranolazine
- No additional medication (No Intervention): No additional medication - control group

INTERVENTIONS:
Drug: Ranolazine — Improvement of myocardial microcirculation
  Other Names: Ranexa
  Arms: Ranolazine

SUMMARY:
The aim of the RIMINI-Trial is to examine the effect of Ranolazine on ischemic myocardium in acute myocardial ischemia.

A pilot-trial by Venkatamaran et al. recently demonstrated, that the area of ischemic myocardium in patients with stable coronary artery disease can be reduced by Ranolazine-treatment2. This effect was shown by significantly reduced areas of atypical or dysfunctional myocardium in SPECT-examinations.

The dimension of myocardial damage (i.e. area of ischemic myocardium) is directly related to the rate of complications (i.e. left-ventricular pump failure, malignant arrhythmia) and the grade of Rehabilitation to daily life (i.e. persistent reduced left-ventricular ejection fraction).

In patients with stable angina pectoris, Ranolazine is used with beneficial results1. Ranolazine improves diastolic blood flow and therefore microcirculation in the myocardium by reducing diastolic tension (via inhibiting late Na+-Influx and consecutive Ca2+-Overload).

Recently published data2 showed that treatment with Ranolazine significantly reduces the ischemic area in chronic damaged myocardium. This is due the effect of improved microcirculation in hibernating myocardium.

Early administration of Ranolazine and improvement of microcirculation in patients with acute damaged myocardium (i.e. directly after acute ischemia) should lead to a recruitment and re-uptake of cardiac activity of hibernating myocardium.

For the RIMINI-Trial patients are given Ranolazine on top of the guideline-based treatment to reduce the area of acute ischemic myocardium.

Patients with unstable angina pectoris and proof of acute cardiac ischemia, proof of myocardial dyskinesia and angina pectoris in the patient history will receive unaltered guideline-based therapy for acute cardiac ischemia5,6. All necessary procedures will be performed to stabilize patients to a hemodynamically compensated state and patients are then transferred to receive cardiac catheterization (angiography and angioplasty if necessary).

After patients are stabilized Ranolazine will be given additionally to guideline based medication.

The measurement of the ischemic myocardial area will be done via three functional echocardiographies with speckle tracking technique10.

A statistical evaluation of ischemic myocardial area before and after treatment with Ranolazine/Placebo will be done after conclusion of the RIMINI-Trial to show the effect of Ranolazine in acute myocardial ischemia.

DETAILED DESCRIPTION:
The aim of the RIMINI-Trial is to examine the effect of Ranolazine on ischemic myocardium in acute myocardial ischemia.

A pilot-trial by Venkatamaran et al. recently demonstrated, that the area of ischemic myocardium in patients with stable coronary artery disease can be reduced by Ranolazine-treatment2. This effect was shown by significantly reduced areas of atypical or dysfunctional myocardium in SPECT-examinations.

The dimension of myocardial damage (i.e. area of ischemic myocardium) is directly related to:

1. Rate of complications (i.e. left-ventricular pump failure, malignant arrhythmia)
2. Grade of Rehabilitation to daily life (i.e. persistent reduced left-ventricular ejection fraction)

Early angioplasty and coronary medication are key factors for preventing complications and ensuring sufficient rehabilitation. This is done to reduce the ischemic area as best as possible.

In patients with stable angina pectoris, Ranolazine is used with beneficial results1. Ranolazine improves diastolic blood flow and therefore microcirculation in the myocardium by reducing diastolic tension (via inhibiting late Na+-Influx and consecutive Ca2+-Overload).

Recently published data2 showed that treatment with Ranolazine significantly reduces the ischemic area in chronic damaged myocardium. This is due the effect of improved microcirculation in hibernating myocardium.

Early administration of Ranolazine and improvement of microcirculation in patients with acute damaged myocardium (i.e. directly after acute ischemia) should lead to a recruitment and re-uptake of cardiac activity of hibernating myocardium.

For the RIMINI-Trial patients are given Ranolazine on top of the guideline-based treatment to reduce the area of acute ischemic myocardium.

Patients with unstable angina pectoris and proof of acute cardiac ischemia (Serum levels of Troponin-T-hs >14 pg/ml), proof of myocardial dyskinesia and angina pectoris >/=CCS II (Canadian Cardiovascular Society Classification of Angina Pectoris) in the patient history will receive unaltered guideline-based therapy for acute cardiac ischemia5,6. All necessary procedures will be performed to stabilize patients to a hemodynamically compensated state (normalized levels of blood pressure, heart rate, absent malignant arrhythmia, dyspnoea and angina-like symptoms), and patients are then transferred to receive cardiac catheterization (angiography and angioplasty if necessary).

After patients are stabilized (i.e. via angioplasty, medical treatment) Ranolazine will be given additionally to guideline-based medication (Beta-Blocker, ACE-Inhibitor or AT1-Inhibitor, ASS, Clopidogrel, Statins).

The measurement of the ischemic myocardial area will be done via three functional echocardiographies with speckle tracking technique10 (speckle -tracking echocardiography, SPE):

1. The first speckle tracking for screening and will be done directly with patients presenting in the emergency room.
2. After stabilization and coronary angiography or -plasty and before the first dose of Ranolazine is given, the second speckle tracking will be done for baseline.
3. After 42 days of Ranolazine-treatment the third and final speckle tracking echocardiography will be done.

A statistical evaluation of ischemic myocardial area before and after treatment with Ranolazine/Placebo will be done after conclusion of the RIMINI-Trial to show the effect of Ranolazine in acute myocardial ischemia.

For controlling and comparing the effect, the RIMINI-Trial will be single-blinded and compared to a group of patients not treated with Ranolazine. Participants will be randomized to the treatment-group or the no-treatment-group using a computer based randomization-method.

ELIGIBILITY:
Inclusion Criteria:

* Proof of acute cardiac ischemia by elevated serum Troponin T-hs levels > 14 pg/nl
* Proof of myocardial dyskinesia with functional echocardiography ("speckle tracking")
* Stable angina pectoris >/= CCS II in patient history
* Stabilized (i.e. normalized vital parameters) patients after coronary angioplasty or angiography
* Coronary angioplasty or angiography not older than 24 hours
* Written informed consent
* Established standard therapy for coronary artery disease (i.e. Beta-Blocker, ACE-Inhibitor or AT1-Inhibitor, ASS, Clopidogrel, Statins)

Exclusion Criteria:

* Patients younger than 18 years of age
* Acute cardio-pulmonary decompensation
* Middle and high grade liver insufficiency (Child-Pugh Score B and C)
* High grade renal insufficiency (Creatinine-Clearance < 30 ml/min)
* Concomitant treatment with potent inhibitors of CYP3A4
* Concomitant administration of class Ia (e.g. quinidine) or class III (e.g. dofetilide, sotalol) antiarrhythmics, except for amiodarone
* Concomitant administration of > 20 mg simvastatin/day
* Patients with heart failure classification NYHA III and NYHA IV
* Homeless patients and drug-addicted patients
* Pregnant and/or breast-feeding women
* Treatment with Ranolazine prior to enrolment in RIMINI-Trial
* Allergy against Ranolazine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Blankenberg, Prof. Dr., Principal Investigator — Director of University Heart Center Hamburg Eppendorf
Locations (1):
- University Heart Center Hamburg Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Morrow DA, Scirica BM, Karwatowska-Prokopczuk E, Murphy SA, Budaj A, Varshavsky S, Wolff AA, Skene A, McCabe CH, Braunwald E; MERLIN-TIMI 36 Trial Investigators. Effects of ranolazine on recurrent cardiovascular events in patients with non-ST-elevation acute coronary syndromes: the MERLIN-TIMI 36 randomized trial. JAMA. 2007 Apr 25;297(16):1775-83. doi: 10.1001/jama.297.16.1775. PMID 17456819
- [Background] Venkataraman R, Belardinelli L, Blackburn B, Heo J, Iskandrian AE. A study of the effects of ranolazine using automated quantitative analysis of serial myocardial perfusion images. JACC Cardiovasc Imaging. 2009 Nov;2(11):1301-9. doi: 10.1016/j.jcmg.2009.09.006. PMID 19909934
- [Background] El-Kadri M, Sharaf-Dabbagh H, Ramsdale D. Role of antiischemic agents in the management of non-ST elevation acute coronary syndrome (NSTE-ACS). Cardiovasc Ther. 2012 Feb;30(1):e16-22. doi: 10.1111/j.1755-5922.2010.00225.x. Epub 2010 Sep 15. PMID 20840192
- [Background] Van de Werf F, Bax J, Betriu A, Blomstrom-Lundqvist C, Crea F, Falk V, Filippatos G, Fox K, Huber K, Kastrati A, Rosengren A, Steg PG, Tubaro M, Verheugt F, Weidinger F, Weis M; ESC Committee for Practice Guidelines (CPG). Management of acute myocardial infarction in patients presenting with persistent ST-segment elevation: the Task Force on the Management of ST-Segment Elevation Acute Myocardial Infarction of the European Society of Cardiology. Eur Heart J. 2008 Dec;29(23):2909-45. doi: 10.1093/eurheartj/ehn416. Epub 2008 Nov 12. No abstract available. PMID 19004841
- [Background] Task Force for Diagnosis and Treatment of Non-ST-Segment Elevation Acute Coronary Syndromes of European Society of Cardiology; Bassand JP, Hamm CW, Ardissino D, Boersma E, Budaj A, Fernandez-Aviles F, Fox KA, Hasdai D, Ohman EM, Wallentin L, Wijns W. Guidelines for the diagnosis and treatment of non-ST-segment elevation acute coronary syndromes. Eur Heart J. 2007 Jul;28(13):1598-660. doi: 10.1093/eurheartj/ehm161. Epub 2007 Jun 14. No abstract available. PMID 17569677
- [Background] Andersen GO, Knudsen EC, Aukrust P, Yndestad A, Oie E, Muller C, Seljeflot I, Ueland T. Elevated serum osteoprotegerin levels measured early after acute ST-elevation myocardial infarction predict final infarct size. Heart. 2011 Mar;97(6):460-5. doi: 10.1136/hrt.2010.206714. Epub 2011 Jan 26. PMID 21270073
- [Background] Lunde K, Solheim S, Aakhus S, Arnesen H, Abdelnoor M, Egeland T, Endresen K, Ilebekk A, Mangschau A, Fjeld JG, Smith HJ, Taraldsrud E, Grogaard HK, Bjornerheim R, Brekke M, Muller C, Hopp E, Ragnarsson A, Brinchmann JE, Forfang K. Intracoronary injection of mononuclear bone marrow cells in acute myocardial infarction. N Engl J Med. 2006 Sep 21;355(12):1199-209. doi: 10.1056/NEJMoa055706. PMID 16990383
- [Background] Miller TD, Gibbons RJ. Measuring myocardium at risk in acute myocardial infarction--a continuing challenge. J Nucl Cardiol. 2010 Oct;17(5):778-80. doi: 10.1007/s12350-010-9278-3. No abstract available. PMID 20717762
- [Background] Geyer H, Caracciolo G, Abe H, Wilansky S, Carerj S, Gentile F, Nesser HJ, Khandheria B, Narula J, Sengupta PP. Assessment of myocardial mechanics using speckle tracking echocardiography: fundamentals and clinical applications. J Am Soc Echocardiogr. 2010 Apr;23(4):351-69; quiz 453-5. doi: 10.1016/j.echo.2010.02.015. PMID 20362924
- [Derived] Schwemer TF, Radziwolek L, Deutscher N, Diermann N, Sehner S, Blankenberg S, Friedrich FW. Effect of Ranolazine on Ischemic Myocardium IN Patients With Acute Cardiac Ischemia (RIMINI-Trial): A Randomized Controlled Pilot Trial. J Cardiovasc Pharmacol Ther. 2019 Jan;24(1):62-69. doi: 10.1177/1074248418784290. Epub 2018 Jun 24. PMID 29938533
- See also: University Heart Center Hamburg Eppendorf — http://www.uhz.de

RESULTS

PARTICIPANT FLOW:
Recruitment Details: first patient enrolled: 05-Aug-2013 last patient finished: 05-Jun-2015
  All patients were enrolled at University Heart Centre Hamburg Eppendorf
Period: Overall Study
Arm/Group | Ranolazine | No Additional Medication
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranolazine | No Additional Medication | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (9) | 72 (7) | 70 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular Global Strain Rate
Description: Relativ acceleration or deceleration (1/s) of left ventricular myocardial sections compared to direct opposite section. The more positive the value, the more simultaneously the movements, the more hemodynamically better.
Time Frame: 42 days after first dose of Ranolazine
Population: Secondary Outcome Measure data was not collected. Initially planned secondary outcome (e.g. cardiac events) was found to interfere with monitoring drug safety
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Ranolazine | No Additional Medication
Number analyzed (Participants) | 10 | 10
percentage of change | 18 (2) | 23 (3)

ADVERSE EVENTS:
Arm/Group | Ranolazine | No Additional Medication
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes